CLINICAL TRIAL: NCT06011018
Title: Comparison of Effects of Mirror Therapy Combined With Neuromuscular Electrical Stimulation or Binaural Beats Stimulation on Cortical Excitability, Heart Rate Variability and Lower Limb Motor Function in Patients With Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20220175
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Healthy Adults
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy; Electric Stimulation

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned treatment groups:
  1. Mirror Therapy
  2. Mirror Therapy + Electrical Stimulation
  3. Mirror Therapy + Binaural Beat
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mirror therapy (Experimental)
  Interventions: Other: Mirror Therapy
- Mirror Therapy + Electrical Stimulation (Experimental)
  Interventions: Other: Mirror Therapy + Electrical Stimulation
- Mirror Therapy + Binaural Beat (Experimental)
  Interventions: Other: Mirror Therapy + Binaural Beat

INTERVENTIONS:
Other: Mirror Therapy — Sitting, mirror place at the midline between the legs. Unaffected leg is placed in front of the mirror and perform ankle dorsiflexion exercises.
  Duration: 5 seconds, Rest: 5 seconds
  Arms: Mirror therapy
Other: Mirror Therapy + Electrical Stimulation — Same as the mirror therapy protocol. Affected leg: electrical stimulation on tibialis anterior muscle. Frequency: 35 Hz, Pulse width: 250µs, Duration: 5 seconds, Rest: 5 seconds.
  Arms: Mirror Therapy + Electrical Stimulation
Other: Mirror Therapy + Binaural Beat — Same as the mirror therapy protocol. Listen to music (pink noise), with 14Hz binaural beat stimulation
  Arms: Mirror Therapy + Binaural Beat

SUMMARY:
This study aims to compare the effects of mirror therapy combined with either neuromuscular electrical stimulation or binaural beat stimulation on post-stroke lower limb motor function recovery. The study also explores the relationship between patients' cortical excitability and motor function improvement.

ELIGIBILITY:
Inclusion Criteria:

1. First occurrence of stroke≧ 6 months
2. Mini-mental state examination≧24
3. Modified Ashworth's scale of ankle muscle ≦3
4. Sit independently≧30 mins
5. Brunnstrom stage ≧3
6. Aged between 20 and 80 years

Exclusion Criteria:

1. Speech impairment
2. Hearing impairment
3. Visual impairment
4. Other orthopedic diseases or nerve damage
5. Complete sensory impairment
6. Pacemaker or metal implants

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer assessment, lower extremity | 10minutes
  The Fugl-Meyer Assessment for lower extremity is a scale used to evaluate motor and functional recovery in patients with conditions like stroke. It measures muscle strength, movement control, coordination, and balance. Scores range from 0 (no movement) to 34 (full recovery). Higher scores indicate better recovery.

SECONDARY OUTCOMES:
Modified ashworth scale | 5minutes
  The Modified Ashworth Scale assesses muscle spasticity in conditions like stroke or cerebral palsy. Scores range from 0 to 4 or 5, indicating the severity of muscle resistance during passive movement. Higher scores mean more severe spasticity. It guides treatment and tracks progress.
Timed up and go test | 5minutes
  The Timed Up and Go (TUG) test assesses mobility by measuring the time it takes for someone to stand, walk a short distance, turn, and sit back down. Faster times suggest better mobility, while longer times may indicate mobility limitations or fall risk. It's a useful tool to evaluate functional capacity and guide interventions for improved mobility.
The postural assessment scale for stroke patients | 10 minutes
  Higher scores on the Postural Assessment Scale for Stroke Patients (PASS) indicate greater difficulty in postural control and stability after a stroke.
Barthel index | 5minutes
  The Barthel Index assesses a person's ability to independently perform daily activities. Scores range from 0 to 100, with higher scores indicating greater independence.

OTHER OUTCOMES:
Electroencephalography | 20minutes
  Electroencephalography is used obtain power data of total μ (8-12Hz), lower μ (8-10Hz), and upper μ (10-12Hz).
  μ suppression→ a negative value (<0) indicates inhibition of μ waves, indicating activation in the motor cortex(Bae et al., 2012).

CONTACTS AND LOCATIONS:
Overall Officials: LIN JAU HONG, Ph.D., Study Chair — Kaohsiung Medical University,department of Physical Therapy
Locations (1):
- Kaohsiung Medical University, Department of Physical Therapy, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
During the study period, to ensure subject privacy, only the implementers of this research project, monitors, regulatory authorities, and the institutional review board of our institution have the authority to access the data